CLINICAL TRIAL: NCT06832488
Title: A Randomised Control Trial Exploring the Effect of Food Textures on Food Intake and Eating Rate in Care Home Dwelling Older Adults.
Brief Title: Food Texture, Eating Rate and Food Intake in Care Home Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Lisa Methven, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRAS 346597
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition
Keywords: Older adults; Food intake; Food texture; Eating rate; Care homes; Appetite
MeSH Terms: conditions — Malnutrition | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day 1 receiving easier to eat food textures and day 8 receiving more difficult to eat textures (Active Comparator): In this arm participants will receive in the first intervention day the easier to eat food textures and in the second (day 8 after washout) the more difficult to eat food textures
  Interventions: Behavioral: Diet
- Day 1 receiving more difficult to eat food textures and day 8 receiving easier to eat textures (Active Comparator): In this arm participants will receive in the first intervention day the more difficult to eat food textures and in the second (day 8 after washout) the easier to eat food textures
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — To compare the total food and energy intake of the diet with textures that require reduced oral processing versus the diet with textures that require increased oral processing by measuring weight before and after consumption of each meal and snack

SUMMARY:
It's estimated that around 1 in 10 older adults are malnourished or at risk of malnutrition in the UK. In comparison with the general older adult population, care home residents are more likely to be underweight. Many factors can affect food intake and choices of older adults. The previous studies of this PhD project have shown that 1) older adults who eat slower, consume less food and 2) that there are food textures that are consumed at a significantly faster pace than others. Following these results, this research will specifically aim to test if providing meals including food textures that require reduced oral processing can increase eating rate and total food intake in care home dwelling older adults. The potential benefits of this research is to inform how providing appropriate food textures can increase older adults (dwelling in care homes) eating speed, ease oral processing and consequently improve food intake, which can help towards better overall health and quality of life.

Participants will be asked to take part in two study days, one week apart. On the one day they will consume all meals including textures that require reduced oral processing ("easier" food textures), and on the other day all meals including textures that require increased oral processing ("more difficult" food textures). The meals will be balanced for energy content per portion, and all foods will be within the normal range of foods provided in care homes. The researchers will record food and energy intake from each meal, duration of meal and calculate eating rate of each meal.

The research will be recruiting from care homes around England, who have reviewed and agreed will all parts of the research. Participants who consume a regular diet can be included.

DETAILED DESCRIPTION:
The hypothesis of this study is that consumption of all-meals of a study day with food textures that require reduced oral processing versus food textures that require increased oral processing, would lead to increased total daily food and energy intake in care home older adults. The null hypothesis is that the two study days will no differ in food intake and the alternative hypothesis is that the study day with food textures that require increased oral processing will lead to increased food and energy intake..

Study design: This study includes two study days with a one week washout in between them. In one study day all meals of the day will be provided in "more difficult" to eat textures (a diet with food textures that require increased oral processing). In the other study day all meals of the day will be provided in "easier" to eat textures (a diet with food textures that require reduced oral processing). All meals will be prepared and provided by Apetitio Limited, a food company that specialises in designing and delivering foods for older adults. Some options will be provided by the research team following retail purchase (i.e., biscuits, cakes, bread etc.) All meals, recipes, snacks will be to kept consistent across care homes. The time each participant is starting each meal and the time finishing each meal will be recorded, to calculate total eating time. The weight of the food provided and the weight of the food when finished the meal will also be recorded to calculate food intake, and then using the eating time the eating rate of the meal will be calculated. With residents that are able to using rating scales, short questions on appetite, hunger and liking of the meal will be asked before and after each main meal (breakfast, lunch, evening meal). Same snacks and fluid types will be provided in both study days and the snack and fluid intake will be recorded. No other changes in the daily life of the participant will happen. Baseline information from each participant will be collected before the start of the study from the care homes' records.

The above study design and methodology was influenced by previous research that measured eating rate and food intake in similar ways. At the same time, the methods we will use in this study have been selected carefully to be feasible in care homes and minimise effort needed from the participants and carers.

Food/plate waste measurement (in an audit form): To the residents that are not part of the trial, the meals will also be offered as one of the options on each daily menu. From these meals, and in a fully anonymised way, the researchers will collect the total amount of meals leaving the kitchen and the total leftovers/food waste are being thrown away in order to collect the total amount of these meals consumed and the number of the meals. Data will not be identifiable to the individual. These extra data will be collected to support power and study findings, but will not require consent as no individual is participating in the study, this is purely an "audit" of food served and wasted.

The timetable for the stages of the research is as follows: The researchers aim to run the research around spring-summer 2025. Results will be analysed on completion of the study across care homes. Anonymised results will be then published as a scientific paper and will be presented in international conferences (November 2025- May 2026). Results of this study will also be part of the PhD thesis of the student which will be submitted on or before April 2026.

Recruitment will take place initially at a care home level, where the care home manager has reviewed and consented for the care home to participate in the research. Subsequently, care homes' staff will assist with recruiting eligible participants.

The research itself as well as the presence of the researcher in the care home may influence participants behaviour; however this will be consistent in both study days, which will have a week washout period. The randomised order of the study days in each care home will also possibly affect the results; however the researchers will aim to balanced within each care home, if big enough to have more than one units/dining areas and will be considered in the statistical analysis as well.

To define the sample size, power calculations were undertaken through an online power calculator (ClinCalc, 2024), using a two study groups design, continuous primary endpoint, 80% power and alpha <0.05. The calculations, following the primary outcome of the study, were based on previous, published research in free living older adults when compared energy intake in a meal with or without added sauce and found significant differences in the food intake from the meal with sauce(Best and Appleton, 2011). Sample size has been calculated as 28 participants, and accounting for 10% dropouts to 31 participants.

Participants will be approached through the care home staff and will be provided with the participant information leaflet and consent form. If participants don't have capacity to consent, a consultee will be advised and provided the participant information leaflet and consultee consent form

ELIGIBILITY:
Inclusion Criteria:

Care homes:

Care or residential homes, that host older adult residents that are not in end-of-life care or have solely nursing needs

Participants:

* Aged 65+
* Permanent care home residents, living in the care home for at least one month
* Able to provide consent or if not having capacity to consent to have a consultee that can provide consent (noting that residents without capacity to consent will be asked for their assent)
* Able to consume a "regular" care home diet
* Not on any special diet (i.e., for dysphagia, kidney disease etc.)
* Able to consume at least 1 meal a day
* Not being critically ill or on end-of-life care
* Not allergic or intolerant or dislike completely any foods or ingredients in the meals provided

Exclusion Criteria:

Care homes:

That solely provide nursing or end-of-life care

Participants:

* Aged <65 years
* Not living in a care home or living in the care home for less than one month
* Not able to provide consent either by themselves or by a consultee
* Under a special diet and/or not able to consume a "regular" care home diet
* Not able to consume at least 1 meal a day
* Being critically ill/end of life care
* Having allergies/intolerances/aversions to ingredients and foods of the meals provided

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Total daily food and energy intake | 1 day for each diet
  To compare the total food and energy intake of the meals with textures that require reduced oral processing (day with easier to eat textures) versus the meals with textures that require increased oral processing (day with more difficult to eat texts)

SECONDARY OUTCOMES:
Food and energy intake of each meal | Up to 30 minutes for each meal
  To compare the food and energy intake of each meal of the day that have meals with textures that require reduced oral processing versus the days that have meals with textures that require increased oral processing.
Eating rate | Up to 30 minutes for each meal
  To compare the eating rate of the meals with textures that require reduced oral processing versus the meals with textures that require increased oral processing.
Self-reported appetite and meal liking ratings | 2 minutes before and 2 minutes after each meal
  (Where applicable) To assess and compare the self-reported ratings of appetite, fullness and liking of the meals.
  The decision tree approach will be followed and the questions and answers structure follows the publication of Pouyet et al. 2015, Food Quality and Preference
  A 5-point scale system will be used for answers where (1) is the maximum value and (5) the minimum value
  e.g Asking about HUNGER BEFORE THE MEAL
  1. Are you hungry right now?
  * Yes
  * Moderately (3)
  * No
    1a. If yes, how hungry?
  * Extremely hungry (1)
  * Hungry (2)
    1b. If no, how not hungry?
  * Not hungry (4)
  * Extremely not hungry (5)
    1. Extremely hungry, (2) Moderately hungry (3) Neither hungry nor not hungry (4) Moderately not hungry (5) Extremely not hungry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pseudoanonymised data or fully anonymised data will be shared with other researchers.